CLINICAL TRIAL: NCT04369365
Title: A Single-blinded, Randomized, Placebo Controlled Phase II Trial of Prophylactic Treatment With Oral Azithromycin Versus Placebo in Cancer Patients Undergoing Antineoplastic Treatment During the Corona Virus Disease 19 (COVID-19) Pandemic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Matthias Preusser (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Matthias Preusser, Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OnCoVID-19 Trial
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: COVID
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Azithromycin (Active Comparator): weekly oral azithromycin 1500mg for a maximum of 8 weeks
  Interventions: Drug: Azithromycin 500 milligram (mg) oral Tablet
- Arm B: Placebo (Placebo Comparator): weekly oral placebo for a maximum of 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin 500 milligram (mg) oral Tablet — weekly oral use
  Arms: Arm A: Azithromycin
Drug: Placebo — weekly oral use
  Arms: Arm B: Placebo

SUMMARY:
Prophylactic treatment in cancer patients undergoing antineoplastic therapy during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer diagnosis
* Ongoing systemic antineoplastic treatment irrespective of application route
* Age ≥ 18 years
* Life expectancy of at least 3 months
* Adequate renal, cardiac and liver function
* Corrected QT time (QTc) ≤ 450 ms
* Eastern Cooperative Oncology Group (ECOG) performance status of < 3
* Capable of understanding the study and giving informed consent
* Negative COVID-19 test at study entry as measured by routine testing

Exclusion Criteria:

* Use of any investigational agent within 28 days prior to study start
* Patients with active opportunistic infections
* Pregnant or lactating women
* Women of childbearing potential and male subjects not willing to use adequate contraception methods during the study period
* Hypersensitivity to azithromycin or other macrolides
* Concurrent medication with ergotamine, theophylline, digitalis
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Cumulative number of severe acute respiratory syndrome corona virus 2 (SARS-COV-2) infections | 12 weeks after initiation of therapy
  assessed by positive polymerase chain reaction (PCR) from routine nasal swabs (performed every 28 days)

SECONDARY OUTCOMES:
Number of severe COVID-19 cases | 12 weeks after initiation of therapy
  defined as combined endpoint of hospitalization rate or death
Severity of COVID-19 cases | 12 weeks after initiation of therapy
  grading as outlined by the world health organization (WHO)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 weeks after initiation of therapy
  significant clinical and laboratory abnormalities according to CTCAE criteria
Number of viral and bacterial infections | 12 weeks after initiation of therapy
  other than COVID-19
Number of participants with azithromycin-resistant bacterial strains in nasal swabs test | 12 weeks after initiation of therapy
  Development of azithromycin-resistant bacterial strains as assessed by nasal swabs test

CONTACTS AND LOCATIONS:
Locations (1):
- AKH Vienna, Department for Internal Medicine I, Oncology, Vienna, Austria

REFERENCES:
- [Derived] Mair MJ, Maj-Hes A, Nussbaumer-Proll A, Puhr R, Christenheit A, Troch M, Puhr HC, Starzer AM, Steindl A, Eberl S, Haslacher H, Perkmann T, Minichsdorfer C, Prager GW, Lamm WW, Berghoff AS, Kiesewetter B, Zeitlinger M, Preusser M, Raderer M. Prophylactic treatment with oral azithromycin in cancer patients during the COVID-19 pandemic (OnCoVID): a randomized, single-blinded, placebo-controlled phase 2 trial. Infect Agent Cancer. 2023 Feb 12;18(1):9. doi: 10.1186/s13027-023-00487-x. PMID 36782325